CLINICAL TRIAL: NCT01206855
Title: Use of MIST Ultrasound Therapy to Minimize Edema, Bruising and Scarring After Cosmetic Surgery Procedures of the Face and Body
Brief Title: Effectiveness Study of MIST Therapy After Cosmetic Surgery Procedures of the Face and Body
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Celleration, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Celleration-NU-01
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Cosmetic Surgery
Keywords: MIST Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SOC Treated Side of Incision (Active Comparator): One side of the incision will be treated with surgeon's standard postoperative care including cleansing, creams, dressings
  Interventions: Other: Standard Postoperative Incision Care
- MIST Treated Side of Incision (Active Comparator): One half of the incision will receive MIST Therapy treatments 3 times per week for 2 weeks
  Interventions: Device: MIST Therapy

INTERVENTIONS:
Device: MIST Therapy — Low-frequency, non-contact ultrasound system delivering therapeutic ultrasound via a fine saline mist to the wound bed without direct contact of the device with the body.
  Other Names: MIST device; MIST ultrasound treatment
  Arms: MIST Treated Side of Incision
Other: Standard Postoperative Incision Care — Incision cleansing, topical creams, and dressing as needed
  Arms: SOC Treated Side of Incision

SUMMARY:
A clinical trial to evaluate the effect of MIST Therapy on outcomes after cosmetic procedures(including facelifts, blepharoplasties, breast augmentations and reductions, mastopexies, and abdominoplasties) traditionally associated with pain, swelling, bruising, and scarring. The study will test the hypothesis that MIST Therapy can decrease the incidence and severity of these surgical sequelae throughout the acute and sub-acute phases of healing.

DETAILED DESCRIPTION:
A post-market, single-center, prospective, randomized, single-blinded study.

Each subject serves as her/his own control. The procedures chosen are bilateral, and each subject will have one side of the surgical site treated with MIST Therapy and the other side left untreated except for the surgeon's usual postoperative care protocol.

Study objectives: Comparison between MIST-treated side versus the contralateral untreated side on the reduction in swelling, bruising, firmness, pain, and wound healing complications; the potential improvements in scarring; and the improvements in patient satisfaction.

Subject recruitment: A total of 30 subjects will be enrolled into the study. The MIST-treated side will be randomly assigned. The assigned MIST-treated side will be known to the subject and assistant providing MIST Therapy, but will not be known to the Investigator/assessor.

Protocol and procedures: Subjects will be followed until 12 weeks post-surgery. The side assigned for MIST Therapy treatment will be treated weekly, beginning 2-3 days post-surgery, and continuing until 3 weeks post-surgery. A baseline evaluation will include demographic data, medical and surgical history, smoking history, laboratory tests, and digital photography of each side of the wound.

Subjects will be assessed at the following timepoints post-surgery: Days 2,7,14, 21, 28, 42 and 84.

The following procedures and assessments will be obtained at specific timepoints:

* MIST Therapy treatments to the assigned wound side (Days 2, 7, 14, 21)
* Digital photographs (Baseline, Days 14, 21, 42, 84)
* Bruising assessment (Days 7 and 14)
* Pain assessment (Days 7 and 14)
* Swelling assessment (Days 7 and 14)
* Firmness assessment (Days 21 and 42)
* Scar assessment (Days 21 and 84)
* Subject satisfaction (Day 84)
* Concomitant treatments including use of moisturizers, scar creams and compression garments(all timepoints)
* Wound healing complication assessment (all timepoints)
* Adverse event assessment (all timepoints following informed consent)

ELIGIBILITY:
Inclusion Criteria:

* Subject must be between 18-75 years of age
* Subject must be compliant with the study visits
* Subject must be in good health
* Subject must be able to provide written informed consent
* Subject must be undergoing one or more of the following bilateral procedures:

  * Rhytidectomies
  * Blepharoplasty
  * Breast augmentation
  * Mastopexy
  * Breast reduction
  * Abdominoplasty

Exclusion Criteria:

* Subject has any medical condition that would result in poor wound healing
* Subject has any medical condition that would result in poor scarring
* Subject is taking medications that may affect healing or scarring, including Arnica
* Subject has diabetes
* Area to be treated has been irradiated
* Subject is undergoing a secondary procedure that may be associated with prior scar tissue in the area undergoing surgery
* Subject has any medical condition that in the opinion of the Investigator would make the subject an inappropriate candidate for this study, including a higher than usual concern for surgical complications
* Subject has electronic implants or prosthesis
* Subject has cardiac pacemaker
* Pregnant woman
* Skin cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3440 (Actual)
Dates: Start 2010-10; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Reduction in swelling, bruising, firmness and pain | 2-6 weeks
  Outcomes measured by
  * Subject-completed pain and swelling assessments
  * Observer-completed bruising, swelling and firmness assessments
Reduction in wound healing complications | 12 weeks
  Outcome measured by wound evaluations assessing wound dehiscences, suture spitting, and localized wound infections.
Improvements in scarring | 12 weeks
  Outcome measured by Subject-completed and Observer-completed scar assessment scales.

SECONDARY OUTCOMES:
Patient satisfaction | 12 weeks
  Outcome measure: Subject-completed questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Galiano, MD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States